CLINICAL TRIAL: NCT04485143
Title: Cloud-based ECG Monitoring and Healthcare Model Building on the Population With Coronary Artery Revascularization
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Taipei Medical University WanFang Hospital (Other); Taipei Medical University Hospital (Other); Lotung Poh-Ai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N202005037
Record Dates: First submitted 2020-06-29; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Coronary Artery Bypass Graft
Keywords: Percutaneous Coronary Intervention; Coronary Artery Bypass; Phonocardiography, PPG; Bracelet; Vascular Restenosis; Artificial intelligence
MeSH Terms: conditions — Coronary Artery Disease | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: Non-invasive Wearable Device
  Interventions: Device: Wisdom bracelet

INTERVENTIONS:
Device: Wisdom bracelet — routine medical
  Other Names: control group (routine medical)

SUMMARY:
Percutaneous coronary intervention (PCI) and coronary artery bypass graft (CABG) are the golden treatments for stable coronary artery disease (CAD) combined with heart failure (HF). The goal of treating HF patients is to prevent repeated hospitalizations and improve peri-operative survival; clinically, although routines including beta-receptor inhibitors, angiotensin-converting enzyme (ACE) inhibitors, and mineralocorticoids have been shown beneficial for the prognosis, for patients with severely low left ventricular ejection rate, hypotension, and pulmonary disease, the introduction of these drugs in the early postoperative period should still be cautious and may need to be adjusted with related cardiovascular function parameters. Patients with low cardiac output syndrome, ventricular arrhythmia, or hemodynamic instability should be suspected of the failure of bypass grafts if accompanied by changes in the electrocardiogram (EKG) and an increase in myocardial enzymes. Intervention should be carried out as soon as possible after angiography detects graft failure to limit the occurrence of large-scale myocardial injury and prevent the development of severe myocardial failure.

This study is start on June 1 2020. And will include 400 patients who have just undergone PCI and 300 CABG patients who diagnosis of stable coronary artery disease. We will register their medical history, medications, and routine medical examinations within one year, and perform tests such as phonocardiography (Audiocor). They will be worn and measured daily at home after discharge. The data of the electrocardiogram and the PPG bracelet will be registered with their continuous daily values. All subjects tracked the occurrence of adverse medical events within one year after discharge from the hospital. Based on the home-based remote personal care model for patients with CABG, a risk prediction model for heart failure and vascular restenosis was established to effectively reduce medical treatment, adverse events, and medical expenditure.

DETAILED DESCRIPTION:
This study is open, prospective study, multi-center, randomized controlled trial, unobtrusive research. This study is start on June 1 2020. And will include 400 patients who have just undergone PCI and 300 CABG patients who diagnosis of stable coronary artery disease. And random allocation 350 experimental group (Non-invasive Wearable Device) and 350 control group (routine medical).

Ask whether the patients who meet the exclusion criteria are willing to participate in the screening (Screening), if they are willing to join and sign the consent of the subject, and after the patient's condition is stable, conduct an electrocardiogram (V0) before discharge from the hospital. On day 7 (±2 weeks), day 84 (±4 weeks), 168 days (±4 weeks), 252 days (±4 weeks), 336 days (±8 weeks) during routine clinical referral (V1-V5) Both are done once. The results of these two tests and other basic information of the patient, including Demography, Vital Signs, High, Weight, Medication, and European and Taiwan Cardiology Association recommended routine test results of high-risk patients, including Blood Chemistry Panel, NT-proBNP, Echocardiography, Myocardial Perfusion Scan, etc., will record the information of the logged-in subjects on the paper case report form. The CRF only displays the study number, and no subject is available. In addition to the examination of each return visit, the subjects also took the ECG bracelet home at the time of discharge (V0) and wore it every day. After the discharge, the ECG was measured every morning and evening, and their personal activity and sleep were collected. Relevant information. After the subject was discharged from the hospital, the subject tracked the date of all adverse events due to cardiovascular disease within one year, including: heart failure, restenosis due to blood vessel, and non-fatal myocardial infarction , To do blood vessel-related surgery again, and data on the occurrence of death.

ELIGIBILITY:
Inclusion Criteria:

Age>=20,Physician diagnosed with stable coronary artery disease (CAD), accepting PCI patients with stents or CABG, and willing to sign the subject consent and cooperate with return.

Exclusion Criteria:

1. Not eligible
2. Patients judged to be STEMI or NSTEMI by the physician
3. PCI bracket
4. Patients with severe skin damage near the electrode or sensor device.
5. Failure to cooperate in signing consent
6. Those who cannot be admitted to the hospital after the onset and have their first examination before the operation
7. Unable to measure the ECG heart sounds. For example, if you use a heart rate regulator, the ECG will show ventricular tachycardia (VT) and Dextrocardia on admission.
8. Patients who are bedridden and have difficulty in cooperating with return visits
9. Any physician evaluation is not suitable for inclusion in the trial, and subjects who are at high risk in the future cannot cooperate with the follow-up
10. Direct participants in this plan

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age>=20,Physician diagnosed with stable coronary artery disease (CAD), accepting PCI patients with stents or CABG, and willing to sign the subject consent and cooperate with return. And random allocation 350 experimental group (Non-invasive Wearable Device) and 350 control group (routine medical).
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-07-20 (Estimated); Primary Completion 2022-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
death | Within a year
  death, divided into yes or no
Restenosis | Within a year
  Come back to the hospital for PCI or CABG or MI (Judged by the physician) after discharge, divided into yes or no
heart failure | Within a year
  Come back to the hospital for heart failure (Judged by the physician) after discharge, divided into yes or no

SECONDARY OUTCOMES:
heart disease re-hospitalization | Within a year
  Re-hospitalization for heart disease (Judged by the physician) after discharge, divided into yes or no
Stroke re-hospitalization | Within a year
  Re-hospitalization for Stroke (Judged by the physician) after discharge, divided into yes or no
Arrhythmia re-hospitalization | Within a year
  Re-hospitalization for Arrhythmia (Judged by the physician) after discharge, divided into yes or no
Physician adjusts medicine | Within a year
  According to the medicine order issued by the doctor, if there is any adjustment of the medicine, make a record,divided into yes or no
Physician arranges examination early | Within a year
  If the doctor has arranged to do Cardiac ultrasound or stress & redistribution myocardial perfusion scan with SPECT During non-table period, divided into yes or no
Compliance | Within a year
  Judged by the physician, when the patient returns to the consultation, the patient is asked about the compliance with the drug in the past, divided into yes or no
Medical cost | Within a year
  The sum of all medical and health insurance expenses of the patient in the past year

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Chi Liu, MD, Study Chair — Chief, Internal of Medicine

IPD SHARING:
Plan to Share IPD: Undecided